CLINICAL TRIAL: NCT06577675
Title: Progression of a Group of Patients Suffering From Emotional Dysregulation But Heterogeneous in Terms of Diagnosis, Benefiting From the DBT Group Programme.
Acronym: PEAC-TRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20GI281; 2021-A02033-38 (Other: ANSM)
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Emotion Regulation; Emotional Disorder
Keywords: emotional dysregulation; training programme; behaviour therapy; heterogeneous diagnostic groups
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study patients (Experimental): Patients all suffering from emotional dysregulation but heterogeneous in terms of diagnosis and following a group DBT training programme.
  Interventions: Behavioral: Group programme for DBT training

INTERVENTIONS:
Behavioral: Group programme for DBT training — This programme comprises 16 sessions over approximately 5 to 6 months, with one 2.5-hour session every week in a closed group of 8 patients. These sessions will be supervised by two or four carers trained in DBT.

SUMMARY:
Human beings experience emotions and have the ability to manage them, but when these abilities are undermined by mental illness, the result is emotional dysregulation. Borderline patients (1 to 4% of the population) suffer from this symptom and can benefit from a specific therapy: DBT (Dialectical Behaviour Therapy; Linehan, 1993). Created specifically for this condition, DBT significantly reduces emotional dysregulation, a dimension at the root of behavioural disorders that is known to be poorly relieved by drug treatments. The DBT group training programme offers patients the opportunity to learn and practise emotional regulation skills. Four types of skills are taught skills: mindfulness, interpersonal skills, emotional regulation and and distress tolerance. This therapy is part of the psychiatric care, in which patients take responsibility in their own care.

There are many studies showing the effectiveness of DBT and its programme with borderline patients. But there are other pathologies concerned by emotional dysregulation: thymic disorders in particular bipolar (1 to 2.5%), addictive disorders (8 to 10%), eating disorders (ADD, 10%), post-traumatic stress disorder (PTSD, 2%).

DETAILED DESCRIPTION:
A few other studies have demonstrated the efficacy of DBT in patients suffering from other psychiatric disorders (antisocial personality, addictive disorders, particularly alcohol, eating disorders). However, no study has attempted to test the impact of DBT on emotional regulation in a diagnostically heterogeneous group of patients.

The investigators therefore propose, for the first time, to group together different pathologies in the field of emotional regulation disorders (borderline disorders, thymic disorders including bipolarity, anxiety disorders including PTSD, addictive disorders, eating disorders) in order to study the specific influence of the DBT programme on these emotional dysfunctions as its main objective.

The aim of this study is to describe the evolution of a group of diagnostically heterogeneous patients (Borderline Disorder, Bipolar Disorder, Addictive Disorders, CAT Disorders, PTSD) suffering from emotional dysregulation, benefiting from the DBT group programme, in a reduced version of this therapy, since it will take place over 4 to 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated to or entitled under a social security scheme
* Patients aged 18 to 65 suffering from emotional dysregulation and presenting one of the following clinical profiles: borderline disorder, bipolar disorder, addictive disorders, eating disorders, PTSD.
* Follow-up by the Saint Etienne sector (mobile teams, psychological medical centre, intra-hospital services, full-time therapeutic reception centre and day hospitals).
* DERS scale score > 94.
* Patient having received informed information about the study and having signed consent to participate in the study.

Exclusion Criteria:

* Psychotic disorders,
* Melancholic depression,
* Aggressive and hostile behaviour preventing group work,
* Intellectual deficit,
* Patient under guardianship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
DERS (Difficulties in Emotion Regulation Scale) | Weeks 1, 7, 12 and 16
  Measures six dimensions of emotion regulation. The 36 items are scored on a 5-point Likert scale.
  The score is between 36 and 180, 36 for no emotional difficulty and 180 for maximum emotional dysregulation. The higher the score, the greater the difficulty the subject has in emotion regulation.

SECONDARY OUTCOMES:
Quality of life measured by the World Health Organization Quality of Life (WHOQOL-BREF) | Weeks 1 and 16.
  This scale is a 26-item self-questionnaire exploring four domains (physical health, psychological health, social relationships, environment) and two global factors that assess general life satisfaction and sense of personal well-being. Each response is coded on a 5-point Likert scale. The results for each domain give a raw score which, according to the conversion grid, gives a score ranging from 0 to 100 for each domain, with 100 corresponding to a high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yohann MASSE, nurse, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, Saint Priest En Jarez, France

IPD SHARING:
Plan to Share IPD: No